CLINICAL TRIAL: NCT01207115
Title: A Global Multicenter, Randomized, Double-Blind, Placebo- and Active-Controlled Study Comparing the Analgesic Efficacy and Safety of ABT-652 to Placebo in Subjects With Osteoarthritis Pain of the Knee
Brief Title: A Study of ABT-652 in Adults With Osteoarthritis Pain of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-889
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ABT-652 high dose (Experimental): ABT-652 capsules- twice daily for 8 weeks. The dose of ABT-652 will depend on the Arm.
  Interventions: Drug: ABT-652
- ABT-652 low dose (Experimental): ABT-652 capsules - twice daily for 8 weeks. The dose ABT-652 will depend on the Arm
  Interventions: Drug: ABT-652
- Naproxen (Active Comparator): Naproxen capsules- twice daily for 8 weeks
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator): Placebo capsules- twice daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABT-652 — ABT-652 capsules - twice daily for 8 weeks. The dose of ABT-652 will depend on the Arm
  Arms: ABT-652 high dose; ABT-652 low dose
Drug: Placebo — Placebo capsules - twice daily for 8 weeks
  Arms: Placebo
Drug: Naproxen — Naproxen capsules - twice daily for 8 weeks
  Arms: Naproxen

SUMMARY:
To compare the analgesic efficacy and safety of ABT-652 administered twice daily (BID) to placebo in subjects with osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria

* History of OA of the knee joint and meeting American College of Rheumatology (ACR) Clinical and Radiographic criteria,
* Pain score as required by the protocol at Screening and Baseline
* Willing to washout of analgesics and to follow treatment plan, visit schedules and study procedures.

Exclusion Criteria

* History of sensitivity to histamine medications, acetaminophen (paracetamol), or non-steroidal anti-inflammatory drugs (NSAIDs)
* Active gastrointestinal (GI) disease, GI bleeding or GI ulceration, or history of GI bleeding or GI ulceration in the last 6 months
* History of major psychiatric disorders
* Diagnosis of rheumatoid arthritis, autoimmune disorder, arthritis other than osteoarthritis involving the study joint, or other painful syndrome that could interfere with the assessment of pain at the study joint
* Any cardiac, respiratory, neurological or other medical condition or illness that is not well controlled with treatment

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
24-hour average pain score measured by Visual Analog Scale | 8 weeks
  Subject reported pain intensity measured by Visual Analog Scale (0-100)

SECONDARY OUTCOMES:
Western Ontario and McMaster (WOMAC™ ) Osteoarthritis subscales, Pain, Physical Function and Stiffness scores | 8 weeks
  Self administered, patient-centered, health status questionnaire
Subject's Global Assessment of Arthritis Status | 8 weeks
  Subject reported assessment of arthritis status measured by Visual Analogue Scale (0-100)
Brief Pain Inventory | 8 weeks
  Subject reported pain intensity and intereference (scale 0-10)
SF-36v2™ Health Status Survey | 8 weeks
  There is no formal title for this quality of life survey, this is the only name for this measure. Subject reported quality of life survey

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Duan, MD, Study Director — AbbVie
Locations (38):
- United States (23):
  - Site Reference ID/Investigator# 37220, Chandler, Arizona
  - Site Reference ID/Investigator# 37223, Tempe, Arizona
  - Site Reference ID/Investigator# 37215, Tucson, Arizona
  - Site Reference ID/Investigator# 37221, Anaheim, California
  - Site Reference ID/Investigator# 37222, Burbank, California
  - Site Reference ID/Investigator# 35956, Chino, California
  - Site Reference ID/Investigator# 37053, La Mesa, California
  - Site Reference ID/Investigator# 37218, Lomita, California
  - Site Reference ID/Investigator# 37227, Milford, Connecticut
  - Site Reference ID/Investigator# 37229, Boynton Beach, Florida
  - Site Reference ID/Investigator# 37209, Ocala, Florida
  - Site Reference ID/Investigator# 37212, Plantation, Florida
  - Site Reference ID/Investigator# 35961, South Miami, Florida
  - Site Reference ID/Investigator# 37207, Valparaiso, Indiana
  - Site Reference ID/Investigator# 37217, Brooklyn Center, Minnesota
  - Site Reference ID/Investigator# 37228, St Louis, Missouri
  - Site Reference ID/Investigator# 35959, New York, New York
  - Site Reference ID/Investigator# 37211, Salisbury, North Carolina
  - Site Reference ID/Investigator# 37214, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 37205, Wyomissing, Pennsylvania
  - Site Reference ID/Investigator# 37208, Austin, Texas
  - Site Reference ID/Investigator# 37213, San Antonio, Texas
  - Site Reference ID/Investigator# 35953, Richmond, Virginia
- Australia (6):
  - Site Reference ID/Investigator# 41782, Brisbane
  - Site Reference ID/Investigator# 41779, Campsie, Sydney
  - Site Reference ID/Investigator# 41778, Clayton
  - Site Reference ID/Investigator# 41785, Fitzroy
  - Site Reference ID/Investigator# 41582, Kogarah
  - Site Reference ID/Investigator# 41776, Malvern East
- Canada (4):
  - Site Reference ID/Investigator# 41563, Montreal
  - Site Reference ID/Investigator# 41566, Newmarket
  - Site Reference ID/Investigator# 41565, Pointe-Claire
  - Site Reference ID/Investigator# 41562, Sainte-Foy, Quebec
- Site Reference ID/Investigator# 41951, Santiago, Chile
- Puerto Rico (4):
  - Site Reference ID/Investigator# 37183, Caguas
  - Site Reference ID/Investigator# 37622, Ponce
  - Site Reference ID/Investigator# 35966, San Juan
  - Site Reference ID/Investigator# 37184, Trujillo Alto